CLINICAL TRIAL: NCT03052764
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate an Alternative Injection Paradigm for OnabotulinumtoxinA (BOTOX®) in the Treatment of Overactive Bladder in Patients With Urinary Incontinence (LO-BOT)
Brief Title: Evaluation of an Alternative Injection Paradigm for OnabotulinumtoxinA (BOTOX®) in the Treatment of Overactive Bladder in Patients With Urinary Incontinence
Acronym: LO-BOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMO-US-URO-0470
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Urinary Bladder, Overactive; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOTOX® 100 U/BOTOX® 100 U (Active Comparator): BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder on Day 1 and a second injection BOTOX® 100 U after Week 12 if applicable.
  Interventions: Biological: onabotulinumtoxinA
- Placebo/BOTOX® 100 U (Placebo Comparator): Placebo (saline) injection into the bladder on Day 1 and a second injection BOTOX® 100 U after Week 12 if applicable.
  Interventions: Biological: onabotulinumtoxinA; Drug: Placebo (saline)

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA (BOTOX®) injection into the bladder.
  Other Names: BOTOX®; botulinum toxin Type A
Drug: Placebo (saline) — Placebo (saline) injection into the bladder.
  Arms: Placebo/BOTOX® 100 U

SUMMARY:
This study will evaluate the efficacy and safety of onabotulinumtoxinA 100 U (BOTOX®), compared to placebo, when injected into the bladder using an alternative injection paradigm in reducing the number of daily urinary incontinence episodes in patients with overactive bladder (OAB) and urinary incontinence whose symptoms have not been adequately managed with an anticholinergic.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs ≥ 40 kg (88 lb)
* Participant has symptoms of Over Active Bladder (OAB) (frequency and urgency) with urinary incontinence for a period of at least 6 months immediately prior to screening.

Exclusion Criteria:

* Participant has symptoms of OAB due to any known neurological reason (eg, spinal cord injury, multiple sclerosis, cerebrovascular accident, Alzheimer's disease, Parkinson's disease, etc.)
* Participant has received pharmacologic therapy to treat symptoms of OAB, including nocturia, within 7 days of the start of the screening period procedures
* Participant uses clean intermittent catheterization (CIC) or indwelling catheter to manage urinary incontinence
* Participant has been treated with any intravesical pharmacologic agent (eg, capsaicin, resiniferatoxin) within 12 months of Day 1
* Participant has had previous or current botulinum toxin therapy of any serotype for any urological condition
* Participant has had previous or current botulinum toxin therapy of any serotype for any non-urological condition within 12 weeks of Day 1
* Participant has been immunized for any botulinum toxin serotype
* Participant has history or evidence of any pelvic or urological abnormalities, bladder surgery or disease, other than OAB, that may affect bladder function
* Participant has an active genital infection, other than genital warts, either concurrently or within 4 weeks prior to screening
* Participant has a history or current diagnosis of bladder cancer or other urothelial malignancy
* Participant is male with previous or current diagnosis of prostate cancer
* Participant has a history of 2 or more urinary tract infections (UTIs) within 6 months of Day 1 or is taking prophylactic antibiotics to prevent chronic UTIs
* Participant has current or previous uninvestigated hematuria
* Participant has hemophilia, or other clotting factor deficiencies, or disorders that cause bleeding diathesis
* Participant cannot withhold any antiplatelet, anticoagulant therapy or medications with anticoagulant effects for 3 days prior to Day 1
* Participant has a known allergy or sensitivity to any botulinum toxin preparation
* Participant has any medical condition that may put him/her at increased risk with exposure to BOTOX® including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Participant has current swallowing or breathing difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Fetterolf, Study Director — Allergan; Amin Boroujerdi, Study Director — Allergan
Locations (31):
- United States (31):
  - Orange County Urology Associates, Laguna Hills, California
  - Tower Urology, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - PMG Research of Christie Clinic, Champaign, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Women's Health Advantage, Fort Wayne, Indiana
  - Urogynecology Associates, Indianapolis, Indiana
  - Urology of Indiana, Noblesville, Indiana
  - Iowa Clinic, West Des Moines, Iowa
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology, Owings Mills, Maryland
  - Beyer Research, Kalamazoo, Michigan
  - Michigan Institute of Urology, P.C., Troy, Michigan
  - Adult and Pediatric Urology, Omaha, Nebraska
  - Premier Urology LLC, Edison, New Jersey
  - Western New York Urology Associates, Cheektowaga, New York
  - Manhattan Medical Research, New York, New York
  - Advanced Urology Centers of NY A division of IMP, Plainview, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Sandhills Medical Center, Hamlet, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Center for Pelvic Health, Franklin, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Virginia Urology, Richmond, Virginia
  - Virginia Urology Center, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington

REFERENCES:
- [Derived] Poster. Female Pelvic Med Reconstr Surg. 2020 Oct 1;26(10S Suppl 1):S89-S189. doi: 10.1097/SPV.0000000000000936. No abstract available. PMID 33955921
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- BOTOX® 100 U/BOTOX® 100 U: BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder on Day 1 in the Double-Blind Treatment Period and a second injection BOTOX® 100 U after Week 12 if applicable in the Open-Label Re-Treatment Period.
- Placebo/BOTOX® 100 U: Placebo (saline) injection into the bladder on Day 1 in the Double-Blind Treatment Period and a second injection BOTOX® 100 U after Week 12 if applicable in the Open-Label Re-Treatment Period.
Period: Double-Blind Treatment Period
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Started | 80 | 40
mITT | 78 | 39
Completed | 70 | 37
Not Completed | 10 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Reason not Specified | 2 | 1
Period: Open-Label Re-Treatment Period
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Started | 58 | 33
Completed | 58 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U | Total
Number analyzed (Participants) | 80 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.91) | 61.9 (11.26) | 61.0 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 40 | 115
  Male | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 65 | 39 | 104
  Black | 9 | 1 | 10
  Asian | 3 | 0 | 3
  Other | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 75 | 38 | 113
  Hispanic or Latino | 5 | 2 | 7
Daily Average Number of Urinary Incontinence Episodes [Mean (Standard Deviation); unit: incontinence episodes per day] — The participant recorded urinary incontinence in a 3-day bladder diary. Data for the three days was averaged. Population: Modified Intent-to-treat (mITT) Population included all randomized participants who had at least one efficacy assessment at Baseline and a postbaseline visit.
  incontinence episodes per day
    number analyzed (Participants) | 78 | 39 | 117
    (all) | 6.31 (4.341) | 6.34 (3.061) | 6.32 (3.947)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Number of Urinary Incontinence Episodes
Description: The participant recorded urinary incontinence in a 3-day bladder diary. Data for the three days was averaged. A negative change from Baseline indicates improvement. An analysis of covariance (ANCOVA) model with treatment as a factor at 2 levels, and the number of Urgency Urinary Incontinence (UUI) episodes reported at Baseline (<= 9 versus > 9 daily episodes) and Baseline daily average number of episodes of incontinence as covariates was used for analyses.
Time Frame: Baseline (3 consecutive days during the Screening Period; within 35 days prior to Day 1) to 3 consecutive days prior to Week 12
Population: Modified Intent-to-treat (mITT) Population included all randomized participants who had at least one efficacy assessment at Baseline and a postbaseline visit.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes per day
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 78 | 39
incontinence episodes per day | -2.99 (0.488) | -0.42 (0.612)
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; p < .0001, ANCOVA; Least Squares Mean Difference = -2.57, 95% CI 2-sided [-3.68 to -1.46], Standard Error of Mean 0.561

2. Secondary Outcome: Percentage of Participants Who Achieved Complete Continence
Description: Complete continence is defined as 100% reduction in urinary incontinence from Baseline.
Time Frame: Baseline (3 consecutive days during the Screening Period; within 35 days prior to Day 1) to 3 consecutive days prior to Week 12]
Population: mITT Population included all randomized participants who had at least one efficacy assessment at Baseline and a postbaseline visit. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 72 | 37
percentage of participants | 13.9 | 2.7
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; Odds Ratio (OR) = 6.15, 95% CI 2-sided [0.75 to 50.37] — Values obtained were from a Cochran Mantel-Haenszel test adjusting for the number of UUI episodes reported at Baseline (<= 9 versus > 9 daily episodes)at each scheduled visit

3. Secondary Outcome: Change From Baseline in Daily Average Number of Micturition Episodes
Description: The participant recorded the number of micturition episodes in a 3-day bladder diary. Data for the three days was averaged. A negative change from Baseline indicates improvement. An ANCOVA model with treatment as a factor at 2 levels, and the number of UUI episodes reported at Baseline (<= 9 versus > 9 daily episodes) and Baseline daily average number of micturition as covariates was used for analyses.
Time Frame: as for outcome 1
Population: mITT Population included all randomized participants who had at least one efficacy assessment at Baseline and a postbaseline visit. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: micturition episodes per day
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 72 | 37
micturition episodes per day | -2.25 (0.421) | -0.01 (0.525)
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; p < .0001, ANCOVA; Least Squares Mean Difference = -2.24, 95% CI 2-sided [-3.30 to -1.18], Standard Error of Mean 0.534

4. Secondary Outcome: Change From Baseline in Daily Average Number of Urgency Episodes
Description: The participant recorded the number of urgency episode in a 3-day bladder diary. Data for the three days was averaged. A negative change from Baseline indicates improvement. An ANCOVA model with treatment as a factor at 2 levels, and the number of UUI episodes reported at Baseline (<= 9 versus > 9 daily episodes) and Baseline daily average number of urgency episodes as covariates was used for analyses.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: urgency episodes per day
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 72 | 37
urgency episodes per day | -2.79 (0.491) | -0.23 (0.618)
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; p < .0001, ANCOVA; Least Squares Mean Difference = -2.56, 95% CI 2-sided [-3.73 to -1.39], Standard Error of Mean 0.590

5. Secondary Outcome: Change From Baseline in Daily Average Number of Nocturia Episodes
Description: The participants recorded the number of nocturia episodes in a 3-day bladder diary. Data for the three days was averaged. A negative change from Baseline indicates improvement. An ANCOVA model with treatment as a factor at 2 levels, and the number of UUI episodes reported at Baseline (<= 9 versus > 9 daily episodes) and Baseline daily average number of nocturia episodes as covariates was used for analyses.
Time Frame: Baseline (3 consecutive days during the Screening Period; within 35 days prior to Day 1) to, 3 consecutive days prior to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes per day
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 72 | 37
nocturia episodes per day | -0.53 (0.154) | 0.17 (0.193)
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; p = 0.0004, ANCOVA; Least Squares Mean Difference = -0.71, 95% CI 2-sided [-1.09 to -0.32], Standard Error of Mean 0.192

6. Secondary Outcome: Percentage of Participants Who Have a Positive Treatment Response on the Treatment Benefit Scale (TBS)
Description: The participant rated their condition during treatment using the TBS 4-point scale where: 1=greatly improved, 2=improved, 3=not changed or 4=worsened. A positive treatment response is either as score of 1=greatly improved or 2=improved.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX® 100 U/BOTOX® 100 U | Placebo/BOTOX® 100 U
Number analyzed (Participants) | 50 | 17
percentage of participants | 74.0 | 17.6
Statistical Analysis 1: Comparison: BOTOX® 100 U/BOTOX® 100 U vs Placebo/BOTOX® 100 U; Test type: Superiority; Odds Ratio (OR) = 13.03, 95% CI 2-sided [3.23 to 52.57] — Values were obtained from a Cochran Mantel-Haenszel test adjusting for the number of UUI episodes reported at Baseline (<= 9 versus > 9 daily episodes) at each scheduled visit

ADVERSE EVENTS:
Time Frame: Randomization to the Study Exit Visit (Up to 70 Weeks)
Description: ITT population, all randomized participants, was used to determine the number at risk for All-Cause Mortality. Safety Population, all participants who received study drug, was used to determine the number of participants at risk for Adverse Events.
Groups:
- Double Blind: BOTOX® 100 U: BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder on Day 1 in the Double-Blind Treatment Period.
- Double Blind: Placebo: Placebo (saline) injection into the bladder on Day 1 in the Double-Blind Treatment Period.
- Open Label: BOTOX® 100 U/BOTOX® 100 U: BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder in the Open-Label Re-Treatment Period in participants who previously received BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder on Day 1.
- Open Label: Placebo/BOTOX® 100 U: BOTOX® (onabotulinumtoxinA) 100 U injection into the bladder in the Open-Label Re-Treatment Period in participants who previously received Placebo (saline) injection into the bladder on Day 1.
Arm/Group | Double Blind: BOTOX® 100 U | Double Blind: Placebo | Open Label: BOTOX® 100 U/BOTOX® 100 U | Open Label: Placebo/BOTOX® 100 U
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/40 | 0/58 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/78 | 2/39 | 2/58 | 1/33
Other Adverse Events (participants affected / at risk) | 31/78 | 13/39 | 14/58 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: BOTOX® 100 U (N=78) | Double Blind: Placebo (N=39) | Open Label: BOTOX® 100 U/BOTOX® 100 U (N=58) | Open Label: Placebo/BOTOX® 100 U (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: BOTOX® 100 U (N=78) | Double Blind: Placebo (N=39) | Open Label: BOTOX® 100 U/BOTOX® 100 U (N=58) | Open Label: Placebo/BOTOX® 100 U (N=33)
Dysuria (Renal and urinary disorders) | 4 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 28 | 11 | 14 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03052764/SAP_000.pdf
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT03052764/Prot_001.pdf